CLINICAL TRIAL: NCT05759273
Title: Retrospective, Noninterventional Study Assessing the Real-Life Use of The Long-Acting 6-Month Triptorelin Formulation as A Treatment for Different Stages of Prostate Cancer in Italy - REAL6T
Brief Title: A Study to Observe Demography and the Outcome of Prostate Cancer Patients Treated With 6-month Triptorelin Formulation in Italy
Acronym: REAL6T
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52014-454
Record Dates: First submitted 2023-02-17; First posted 2023-03-08 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Triptorelin 6 Month Formulation: Participants treated with the 6-month triptorelin formulation

SUMMARY:
The participants of this study had Prostate Cancer. Prostate cancer is cancer that occurs in the prostate, a small gland in the male reproductive system. This study will collect data on the use of the 6-month triptorelin formulation (Decapeptyl®) in local routine clinical practice as a treatment for different stages of prostate cancer. The aim of this study will be to describe participant characteristics, as well as disease and treatment characteristics before the first injection with the 6-month triptorelin formulation in Italy. The decision to prescribe this product and all hospital visits, dose adjustments, assessments and procedures were made according to routine clinical practice at the time and independently of the decision to enroll the participants in this data collection study.

ELIGIBILITY:
Inclusion Criteria :

* Participants must have a documented diagnosis of prostate cancer, as per the following disease status groups: - participants with intermediate risk prostate cancer with indication to radiotherapy treated with neoadjuvant and concomitant hormonal therapy; - participants with high risk prostate cancer after radical prostatectomy or radiotherapy, treated with adjuvant hormonal therapy; - participants with advanced/metastatic prostate cancer treated with long-term hormonal therapy; - participants treated with primary therapy (i.e. surgery or radiotherapy) with biochemical recurrence; - participants with castration-resistant prostate cancer;
* Participants must have received a minimum of one injection with the 6 month triptorelin formulation according to this product's local label, during the participant identification period;
* Participants must have a minimum of 6 months of follow-up data recorded on their medical files after the first injection with the 6-month formulation, and until death or 06 July 2022, whichever comes first;
* Participants may have received previous treatment with an LHRH analogue;
* Participants must have at least one document analysis of PSA levels recorded before the injection with the 6-month formulation;
* Participants with castration status achieved with any LHRH analogue who switched to the 6-month triptorelin formulation must have a minimum of two documented analysis of testosterone levels: (a) one performed before the first ever injection with the 6-month formulation, if available, and one performed during the period covered by treatment with this formulation to confirm castration maintenance in the participant SMD form protocol master data-OBS / Version 1 OR (b) both analyses performed during the period covered by treatment with this formulation;
* Noncastrated participants or castration-naïve participants must have a minimum of two documented analysis of testosterone levels: (a) one performed before the first ever injection with the 6-month formulation, if available, and one performed during the period covered by the treatment with this formulation to confirm that castration status has been reached; OR (b) both analyses performed during the period covered by treatment with this formulation. Note: if available, another testosterone analysis performed during the period covered by the treatment with this formulation will also be collected to confirm that castration status was maintained in the participant; Note: A noncastrated participant is defined as a participant who was not receiving any testosterone-blocking treatment at the time of the first injection with the 6-month triptorelin formulation but had history of previous ADT agents. A castration-naïve participant is defined as a participant that never received any testosterone-blocking treatment prior to the first injection with the 6-month formulation.
* Provision of written ICF to the extent required according to applicable national local regulations for a retrospective, noninterventional study;

Exclusion Criteria :

* Have missing PSA data before having received the first injection with the 6 month triptorelin formulation;
* Were diagnosed with low-risk or localised prostate cancer;
* Do not fulfil all the inclusion criteria.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is planned to include participants with different stages of prostate cancer excluding low risks and localised prostate cancer, in whom a decision to treat with the 6-month triptorelin formulation had been made before the start of this study and as guided by Italy's label for Decapeptyl®. Eligible participants may or may not have had previous treatment with other LHRH analogues and triptorelin formulations except the 6-month triptorelin formulation.
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Naive to Androgen Deprivation Therapy (ADT), Non-naive to ADT and Castrated | Before first Injection (before day 1)
Demographic Characteristic: Age of Participants | Before first Injection (before day 1)
  The age of study participants will be reported.
Demographic Characteristic: Body Mass Index (BMI) | Before first Injection (before day 1)
  BMI of study participants will be reported.
Testosterone Levels | Before first Injection (before day 1)
  Participants serum testosterone levels will be assessed.
Tumor Characteristics as Evaluated by Eastern Cooperative Oncology Group (ECOG) Score | Before first Injection (before day 1)
  Tumor characteristics, collected by ECOG Score at the nearest visit just before the injection.
Tumor Characteristics as Evaluated by Tumor Node Metastasis (TNM) Staging System | Before first Injection (before day 1)
  Tumor characteristics, collected by TNM staging system at the nearest visit just before the injection.
Tumor Characteristics as Evaluated by Grade Group and/or Gleason Score | Before first Injection (before day 1)
  Tumor characteristics, collected by Grade Group and/or Gleason Score at the nearest visit just before the injection.
Prostate Cancer-specific Antigen(PSA) Levels | Before first Injection (before day 1)
Describe Data of Participants with Prostate Cancer History | Before first Injection (before day 1)
  Describe Data including primary treatment or active surveillance, and other therapies.

SECONDARY OUTCOMES:
Reasons for Choosing the 6-month Triptorelin Formulation | From first injection (Day 1) with the 6-month formulation up to 6 months after the last injection with this product
Percentage of Participants who Either Permanently or Temporarily Discontinued 6-month Triptorelin Formulation | From first injection (Day 1) with the 6-month formulation up to 6 months after the last injection with this product
Duration of Treatment with 6-month Triptorelin Formulation | From first injection (Day 1) with the 6-month formulation up to 6 months after the last injection with this product
Percentage of Participants whose Serum Testosterone Levels Presented Castration Levels (testosterone levels <50 nanograms per deciliter) | From first injection (Day 1) with the 6-month formulation up to 6 months after the last injection with this product
Percentage of Participants Using Prostate Cancer-related Concomitant Therapies | From first injection (Day 1) with the 6-month formulation up to 6 months after the last injection with this product
  Concomitant therapies are defined such as combined treatments (chemotherapy and/or androgen receptor targeted agents (ARTAs; enzalutamide, abiraterone, etc.) and/or radiotherapy.
Prostate Cancer-specific Antigen (PSA) Levels | At first injection (Day 1) with the 6-month triptorelin formulation up to the 6 months after the last injection with this product
Percentage of Participants who Switched to 6-month Triptorelin Formulation From the 3-Month Triptorelin Formulation or Another LHRH Analogue | At first injection (Day 1) with the 6-month triptorelin formulation up to the 6 months after the last injection with this product
  Percentage of participants who switched the treatment along with the reasons for switching the treatment will be reported.
Percentage of Participants who Switched to the 3-month triptorelin Formulation or Another Luteinizing Hormone-releasing Hormone (LHRH) Analogue from 6-month formulation | At first injection (Day 1) with the 6-month triptorelin formulation up to the 6 months after the last injection with this product
  Percentage of participants who switched the treatment along with the reasons for switching the treatment will be reported.
Potential Factors Predictive of any Treatment Switch | At first injection (Day 1) with the 6-month triptorelin formulation up to the 6 months after the last injection with this product
  Potential factors such as PSA levels, prostate cancer aggressiveness criteria (based on tumor histological assessment), age, BMI, physical condition (ECOG scale), comorbidities, etc.) leading to treatment switch will be identified.
Percentage of Participants who Were Noncastrated or Castration-naïve and who Presented Serum Testosterone Levels Corresponding to Castration | Day 45 up to 6 months after the last injection with this product
  Castration is defined as a testosterone level <50 ng/dL among all testosterone evaluations available in the participants' medical files
Percentage of Participants Whose Serum Testosterone Levels Never Reached Castration Levels | During treatment with the 6-month formulation (approximatively three years of existing participants data).
  Castration is defined as a testosterone level <50 ng/dL among all testosterone evaluations available in the participants medical files.
Percentage of Participants With Triptorelin-related Adverse events (AEs), Serious Adverse Events (SAEs), Non-SAEs and as well as Special Situations AEs | From first injection (at day 1) with the 6-month formulation up to 6 months after the last injection with this product.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (13):
- Italy (13):
  - Humanitas Gavazzeni, Bergamo
  - AOU Policlinico "Gaspare Rodolico", Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale ICOT, Latina
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS Ospedale Sacro Cuore-Don Calabria, Cancer Care Center Negrar, Negrar
  - Ospedale Buccheri La Ferla Fatebenefratelli di Palermo, Palermo
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale Santa Maria delle Grazia, Pozzuoli
  - Azienda Ospedaliera Universitaria Sant'Andrea, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Ospedale Sant'Anna, San Fermo della Battaglia
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/